CLINICAL TRIAL: NCT03672292
Title: A Multicenter, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of the Coadministration of SCY-078 With Voriconazole in Patients With Invasive Pulmonary Aspergillosis
Brief Title: Evaluate Safety and Efficacy of the Coadministration of Ibrexafungerp With Voriconazole in Patients With Invasive Pulmonary Aspergillosis
Acronym: SCYNERGIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment took longer than anticipated (slow enrollment during COVID).
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCY-078-206; 2018-002565-18 (EudraCT Number)
Record Dates: First submitted 2018-09-11; First posted 2018-09-14 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Invasive Pulmonary Aspergillosis
Keywords: Aspergillosis; SCY-078; Ibrexafungerp; Coadministration
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; Aspergillosis | interventions — ibrexafungerp; Voriconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SCY-078 plus Voriconazole (Experimental): Either IV voriconazole (loading dose of 6 mg/kg BID on Day 1 followed by maintenance dose of 4 mg/kg BID from Day 2 onwards) OR oral voriconazole (loading dose of 400 mg BID on Day 1 followed by maintenance dose of 200 mg BID from Day 2 onwards).
  PLUS Oral SCY-078 tablets (loading dose of 500 mg BID on Days 1 and 2 followed by maintenance dose of 500 mg QD from Day 3 onwards). Treatment duration = minimum 6 weeks/Max 13 weeks
  Interventions: Drug: SCY-078; Drug: Voriconazole
- Voriconazole mono-therapy (Placebo Comparator): Either IV voriconazole (loading dose of 6 mg/kg BID on Day 1 followed by maintenance dose of 4 mg/kg BID from Day 2 onwards) OR oral voriconazole (loading dose of 400 mg BID on Day 1 followed by maintenance dose of 200 mg BID from Day 2 onwards).
  PLUS Oral Placebo Tablets matching SCY-078 tablets (loading dose of 2 tablets given BID on Days 1 and 2 followed by maintenance dose of 2 tablets given QD from Day 3 onwards).
  Treatment duration = minimum 6 weeks/Max 13 weeks
  Interventions: Drug: Voriconazole; Other: Oral Placebo Tablets

INTERVENTIONS:
Drug: SCY-078 — Oral tablets of SCY-078
  Other Names: Ibrexafungerp
  Arms: SCY-078 plus Voriconazole
Drug: Voriconazole — Voriconazole IV vials or oral tablets
Other: Oral Placebo Tablets — Oral Placebo Tablets matching SCY-078
  Other Names: SCY-078 matching Placebo
  Arms: Voriconazole mono-therapy

SUMMARY:
Study to evaluate the safety and efficacy of coadminstration of SCY-078 with a mold-active azole (voriconazole) compared to voriconazole in patients with invasive pulmonary aspergillosis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, two-arm study to evaluate the safety, tolerability, efficacy and PK of the coadministration of SCY-078 plus voriconazole compared to those of voriconazole in male and female subjects 18 years of age and older with a probable or proven invasive pulmonary aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female adult ≥18 years of age on the day the study informed consent form (ICF) is signed.
2. Subject has a probable or proven IPA based on the protocol-specified criteria (Section 22.3) that requires antifungal treatment. Note: Subjects with possible IPA may enter the screening phase of the study but will only be randomized after meeting criteria for probable or proven IPA.
3. Subject has a result of a serum GMI from a sample obtained within the 96 hours preceding enrollment into the study (Baseline/Treatment Day 1).
4. Subject has a diagnosis of a hematological malignancy or a myelodysplastic syndrome or aplastic anemia or has undergone hematopoietic cell transplantation OR
5. Subject who either recently resolved or ongoing neutropenia (neutropenia defined as absolute neutrophil count < 0.5 x 10⁹/L [< 500/mm³] for > 10 days), temporally related to the onset of fungal disease OR
6. Subject who received treatment with other recognized T-cell immunosuppressants (such as cyclosporine, tacrolimus, monoclonal antibodies or nucleoside analogs) during the past 90 days including solid organ transplant patients OR
7. Subject with inherited severe immunodeficiency (e.g. chronic granulomatous disease, severe combined immunodeficiency)
8. Subject has not received more than 4 days (96 hours) of prior mold-active antifungal therapy for the treatment of the IPA episode in the 7 days preceding enrollment into the study (Baseline/Treatment Day 1). However, subjects who have received more than 4 days but less than 7 days of prior mold-active antifungal therapy for the treatment of the IPA episode in the 7 days preceding enrollment into the study may be enrolled but will require approval from the study medical monitor, who will evaluate each subject on a case-by-case basis.
9. Subject has an IPA episode that, in the investigator´s judgement, requires antifungal therapy and may be adequately treated with voriconazole (i.e., the IPA is not a breakthrough infection while receiving a mold-active azole antifungal [voriconazole, posaconazole, isavuconazole or itraconazole] that requires therapy with a non-azole antifungal agent).

Exclusion Criteria:

1. Subject has a fungal disease with central nervous system involvement suspected at Screening.
2. Subject is receiving, has received or anticipates to be receiving concomitant medications that are listed in the prohibited medication list (Appendix A in full protocol) within the specified washout periods.
3. Subject has a Karnofsky score <20.
4. Subject is expected to die from a non-infectious cause within 30 days from the day the study ICF is signed.
5. Subject is under mechanical ventilation.
6. Subject has abnormal liver test parameters: AST or ALT >5 x ULN and/or total bilirubin >2.5 x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Angulo, MD, Study Director — Scynexis, Inc.
Locations (8):
- United States (3):
  - Brigham Womens Hospital INF 75 Francis Street PBB-A4, Boston, Massachusetts
  - University of Michigan UH south F4005; 1500 E. Medical Center Drive SPC 5378, Ann Arbor, Michigan
  - Wake Forest Baptist Medical Center 1 Medical Center Blvd., Winston-Salem, North Carolina
- Belgium (2):
  - Hematology Department AZ Sint-Jan Brugge - Oostende AV Campus Brugge Ruddershove 10 8000, Bruges
  - UZ Leuven campus Gasthuisberg Hematology Department Herestraat 49 B - 3000, Leuven
- University Health Network at the University of Toronto, Toronto, Ontario, Canada
- Universitaetsklinikum Koeln, Klinisches Studienzentrum 2 für Infektiologie, Klinik I für Innere Medizin Kerpener Str. 62, Bettenhaus Ebene 15 Raum 64, Cologne, Germany
- Alberts Cellular Therapy Center (ACT), Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SCY-078 Plus Voriconazole: Either intravenous (IV) voriconazole (loading dose of 6 milligram/kilogram (mg/kg) twice a day (BID) on Day 1 followed by maintenance dose of 4 mg/kg BID from Day 2 onwards) OR oral voriconazole (loading dose of 400 mg BID on Day 1 followed by maintenance dose of 200 mg BID from Day 2 onwards) PLUS oral SCY-078 tablets (loading dose of 500 mg BID on Days 1 and 2 followed by maintenance dose of 500 mg QD from Day 3 onwards) maximum up to 13 weeks.
- Voriconazole Mono-therapy: Either IV voriconazole (loading dose of 6 mg/kg BID on Day 1 followed by maintenance dose of 4 mg/kg BID from Day 2 onwards) OR oral voriconazole (loading dose of 400 mg BID on Day 1 followed by maintenance dose of 200 mg BID from Day 2 onwards) PLUS Oral Placebo Tablets matching SCY-078 tablets (loading dose of 2 tablets given BID on Days 1 and 2 followed by maintenance dose of 2 tablets given once a day (QD) from Day 3 onwards) maximum up to 13 weeks.
Period: Overall Study
Arm/Group | SCY-078 Plus Voriconazole | Voriconazole Mono-therapy
Started | 10 | 12
Completed | 6 | 8
Not Completed | 4 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCY-078 Plus Voriconazole | Voriconazole Mono-therapy | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.57) | 62.7 (14.08) | 62.2 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 10 | 18
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Drug-related Adverse Events (AEs), Discontinuations Due to AEs and Deaths
Description: Number of participants with treatment-emergent adverse events (TEAEs), drug-related adverse events (AEs), discontinuations due to AEs and deaths.
Time Frame: Up to a maximum of 19 weeks
Population: Safety population including any participant treated with at least one dose of Voriconazole or SCY-078
Measure: Number; unit: participants
Arm/Group | SCY-078 Plus Voriconazole | Voriconazole Mono-therapy
Number analyzed (Participants) | 10 | 12
participants
  Number of participants with treatment emergent adverse events | 10 | 11
  Number of participants with treatment-related adverse events | 4 | 0
  Number of participants discontinued due to adverse event | 2 | 4
  Number of participants who died | 3 | 1

2. Secondary Outcome: Percentage of Participants With Complete Response or Partial Response as Determined by the Data Review Committee (DRC)
Description: Number and percentage of participants with Complete Response or Partial Response as determined by the Data Review Committee (DRC). Complete Response: Survival and resolution of all attributable symptoms and signs of disease; plus, successful radiological outcome; plus, mycological eradication. Partial Response: Survival and partial resolution of attributable symptoms and signs of disease; plus, improvement (at least 25%) of radiological lesions; plus, mycological eradication.
Time Frame: At end of treatment (up to 13 weeks), day 42 and day 84
Population: Intent-to-Treat (ITT) Population including all randomized participants who received at least one dose of randomized study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | SCY-078 Plus Voriconazole | Voriconazole Mono-therapy
Number analyzed (Participants) | 10 | 12
Participants
  Participants with Complete or Partial Response at End of Treatment | 7 | 9
  Participants with Complete or Partial Response at Day 42 | 4 | 6
  Participants with Complete or Partial Response at Day 84 | 4 | 4

3. Secondary Outcome: Percentage of Participants Who Died (Any Cause)
Description: Number and Percentage of participants who died (any cause)
Time Frame: At Day 42 and Day 84
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- SCY-078 and Voriconazole: Either intravenous (IV) voriconazole (loading dose of 6 milligram/kilogram (mg/kg) twice a day (BID) on Day 1 followed by maintenance dose of 4 mg/kg BID from Day 2 onwards) OR oral voriconazole (loading dose of 400 mg BID on Day 1 followed by maintenance dose of 200 mg BID from Day 2 onwards) PLUS oral SCY-078 tablets (loading dose of 500 mg BID on Days 1 and 2 followed by maintenance dose of 500 mg QD from Day 3 onwards) maximum up to 13 weeks.
Arm/Group | SCY-078 and Voriconazole | Voriconazole Mono-Therapy
Number analyzed (Participants) | 10 | 12
Participants
  Day 42 | 1 | 1
  Day 84 | 3 | 1

4. Secondary Outcome: Change in Serum Galactomannan Index (GMI)
Description: Absolute change in serum GMI from from baseline to each time point (Weeks 1, 2, 4 and 6). Negative values indicate a reduction of GMI (i.e., improvement).
Time Frame: Weeks 1, 2, 4 and 6
Population: Participants who have a probable or proven invasive pulmonary aspergillosis at baseline, per DRC, with at least one positive serum GMI at baseline and at least one GMI value at Weeks 1, 2, 4 and/or 6.
Measure: Mean (Full Range); unit: index
Arm/Group | SCY-078 Plus Voriconazole | Voriconazole Mono-therapy
Number analyzed (Participants) | 5 | 5
index
  Week 1 | -0.1870 [-0.790 to 0.130] | -0.4910 [-1.200 to 0.100]
  Week 2: number analyzed (Participants) | 5 | 4
  Week 2 | -0.5240 [-1.680 to 0.280] | -0.4080 [-0.870 to 0.390]
  Week 4: number analyzed (Participants) | 5 | 4
  Week 4 | -0.7500 [-1.880 to 0.000] | -0.9570 [-1.750 to -0.160]
  Week 6: number analyzed (Participants) | 4 | 4
  Week 6 | -0.9950 [-1.900 to -0.030] | -0.9570 [-1.750 to -0.160]

5. Secondary Outcome: Percent of Participants With Changes in GMI
Description: Percentage of participants with the following changes in GMI values from Baseline:
  * Fifty percent reduction or greater at Weeks 1, 2, 4 and 6
  * Twenty-five percent reduction or greater at Weeks 1, 2, 4 and 6
  * Any percent reduction at Weeks 1, 2, 4 and 6
  * Reduction equal to or greater than 0.25 at Weeks 1, 2, 4 and 6
  * Reduction to < 0.5 at Weeks 1, 2, 4 and 6
Time Frame: Weeks 1, 2, 4 and 6 from Baseline
Population: Modified Intent-to-treat (mITT) population including participants who have a probable or proven invasive pulmonary aspergillosis at baseline, per DRC, with at least one positive serum GMI at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | SCY-078 and Voriconazole | Voriconazole Mono-Therapy
Number analyzed (Participants) | 7 | 5
Participants
  Week 1 : Fifty percent reduction or greater | 0 | 1
  Week 1 : Twenty-five percent reduction or greater | 2 | 4
  Week 1 : Any percent reduction | 4 | 4
  Week 1 : Reduction equal to or greater than 0.25 | 2 | 4
  Week 1 : Reduction to < 0.5 | 3 | 2
  Week 2 : Fifty percent reduction or greater | 2 | 2
  Week 2 : Twenty-five percent reduction | 3 | 3
  Week 2 : Any percent reduction | 4 | 3
  Week 2 : Reduction equal to or greater than 0.25 | 3 | 3
  Week 2 : Reduction to < 0.5 | 2 | 1
  Week 4 : Fifty percent reduction or greater | 3 | 3
  Week 4 : Twenty-five percent reduction | 3 | 3
  Week 4 : Any percent reduction | 5 | 3
  Week 4 : Reduction equal to or greater than 0.25 | 3 | 3
  Week 4 : Reduction to < 0.5 | 3 | 0
  Week 6 : Fifty percent reduction or greater | 3 | 3
  Week 6 : Twenty-five percent reduction | 4 | 3
  Week 6 : Any percent reduction | 4 | 4
  Week 6 : Reduction equal to or greater than 0.25 | 3 | 3
  Week 6 : Reduction to < 0.5 | 2 | 1

6. Secondary Outcome: Time to Achieve Serum GMI Change From Baseline
Description: Time (days) to achieve the following changes in serum GMI from Baseline:
  * Fifty percent reduction
  * Twenty-five percent reduction
  * Any percent reduction
  * Reduction equal to or greater than 0.25
Time Frame: Up to a maximum of 19 weeks
Population: Intent-to-treat (ITT) population including participants who have a probable or proven invasive pulmonary aspergillosis at baseline, per DRC.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | SCY-078 and Voriconazole | Voriconazole Mono-Therapy
Number analyzed (Participants) | 10 | 12
Days
  Fifty percent reduction | 28.00 [3.00 to NA] — Insufficient number of participants with events | 29.00 [2.00 to NA] — Insufficient number of participants with events
  Twenty-five percent reduction | 14.00 [3.00 to NA] — Insufficient number of participants with events | 5.50 [2.00 to NA] — Insufficient number of participants with events
  Any percent reduction | 5.00 [3.00 to 9.00] | 3.50 [2.00 to 41.00]
  Reduction equal to or greater than 0.25 | NA [3.00 to NA] — Insufficient number of participants with events | NA [2.00 to NA] — Insufficient number of participants with events

7. Secondary Outcome: Percentage of Participants With a Clinical, Mycological and Radiological Response by DRC
Description: Percentage of participants with:
  * Clinical Response at EoT, Day 42 and Day 84, as determined by the DRC
  * Mycological Response at EoT, Day 42 and Day 84, as determined by the DRC
  * Radiological Response at EoT, Day 42 and Day 84, as determined by the DRC
Time Frame: End of Treatment (EoT), Day 42 and Day 84
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SCY-078 and Voriconazole | Voriconazole Mono-Therapy
Number analyzed (Participants) | 10 | 12
Participants
  Clinical Response at EoT | 6 | 9
  Clinical Response at Day 42 | 4 | 7
  Clinical Response at Day 84 | 3 | 4
  Mycological Response at EoT | 7 | 9
  Mycological Response at Day 42 | 6 | 7
  Mycological Response at Day 84 | 4 | 4
  Radiological Response at EoT | 7 | 9
  Radiological Response at Day 42: number analyzed (Participants) | 6 | 12
  Radiological Response at Day 42 | 5 | 7
  Radiological Response at Day 84 | 4 | 5

8. Secondary Outcome: Percentage of Participants With a Clinical, Mycological and Radiological Response.
Description: Percentage of participants with:
  * Clinical Response at EoT, Day 42 and Day 84, as determined by the Principal Investigator
  * Mycological Response at EoT, Day 42 and Day 84, as determined by the Principal Investigator
  * Radiological Response at EoT, Day 42 and Day 84, as determined by the Principal Investigator
Time Frame: End of Treatment (EoT), Day 42 and Day 84
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SCY-078 and Voriconazole | Voriconazole Mono-Therapy
Number analyzed (Participants) | 10 | 12
Participants
  Clinical Response at EoT | 8 | 10
  Clinical Response at Day 42 | 6 | 9
  Clinical Response at Day 84 | 1 | 0
  Mycological Response at EoT | 7 | 11
  Mycological Response at Day 42 | 6 | 8
  Mycological Response at Day 84 | 1 | 0
  Radiological Response at EoT | 7 | 10
  Radiological Response at Day 42 | 5 | 8
  Radiological Response at Day 84 | 1 | 0

9. Secondary Outcome: SCY-078 and Voriconazole Plasma Concentrations
Description: Voriconazole and SCY-078 plasma concentrations (ng/mL)
Time Frame: Treatment Days 7 and 14 (2-4 hrs post dose)
Population: Participants of study who provide a PK sample
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | SCY-078 and Voriconazole | Voriconazole Mono-Therapy
Number analyzed (Participants) | 9 | 9
nanograms per milliliter (ng/mL)
  Day 7 SCY-078 Concentration: number analyzed (Participants) | 7 | 0
  Day 7 SCY-078 Concentration | 1432.30 (455.59) |
  Day 14 SCY-078 Concentration: number analyzed (Participants) | 6 | 0
  Day 14 SCY-078 Concentration | 1312.03 (422.53) |
  Day 7 Voriconazole Concentration: number analyzed (Participants) | 7 | 8
  Day 7 Voriconazole Concentration | 2609.73 (2060.43) | 2891.72 (1557.20)
  Day 14 Voriconazole Concentration: number analyzed (Participants) | 6 | 8
  Day 14 Voriconazole Concentration | 2074.24 (1201.28) | 2963.49 (1583.51)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 19 weeks
Groups:
- SCY-078 Plus Voriconazole: Either IV voriconazole (loading dose of 6 mg/kg BID on Day 1 followed by maintenance dose of 4 mg/kg BID from Day 2 onwards) OR oral voriconazole (loading dose of 400 mg BID on Day 1 followed by maintenance dose of 200 mg BID from Day 2 onwards).
  PLUS Oral SCY-078 tablets (loading dose of 500 mg BID on Days 1 and 2 followed by maintenance dose of 500 mg QD from Day 3 onwards). Treatment duration = minimum 6 weeks/Max 13 weeks
  SCY-078: Oral tablets of SCY-078
  Voriconazole: Voriconazole IV vials or oral tablets
- Voriconazole Mono-therapy: Either IV voriconazole (loading dose of 6 mg/kg BID on Day 1 followed by maintenance dose of 4 mg/kg BID from Day 2 onwards) OR oral voriconazole (loading dose of 400 mg BID on Day 1 followed by maintenance dose of 200 mg BID from Day 2 onwards).
  PLUS Oral Placebo Tablets matching SCY-078 tablets (loading dose of 2 tablets given BID on Days 1 and 2 followed by maintenance dose of 2 tablets given QD from Day 3 onwards).
  Treatment duration = minimum 6 weeks/Max 13 weeks
  Voriconazole: Voriconazole IV vials or oral tablets
  Oral Placebo Tablets: Oral Placebo Tablets matching SCY-078
Arm/Group | SCY-078 Plus Voriconazole | Voriconazole Mono-therapy
All-Cause Mortality (participants affected / at risk) | 3/10 | 1/12
Serious Adverse Events (participants affected / at risk) | 6/10 | 5/12
Other Adverse Events (participants affected / at risk) | 10/10 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SCY-078 Plus Voriconazole (N=10) | Voriconazole Mono-therapy (N=12)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Acute graft versus host disease in skin (Immune system disorders) | 0 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 2 | 0
Heart transplant rejection (Immune system disorders) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SCY-078 Plus Voriconazole (N=10) | Voriconazole Mono-therapy (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Dry eye (Eye disorders) | 0 | 1
Eye haematoma (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 0
Photopsia (Eye disorders) | 2 | 2
Vision blurred (Eye disorders) | 1 | 1
Visual impairment (Eye disorders) | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Angular cheilitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 1
Oral blood blister (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Terminal ileitis (General disorders) | 1 | 0
Toothache (General disorders) | 1 | 0
Vomiting (General disorders) | 3 | 0
Chest pain (General disorders) | 0 | 2
Disease progression (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 1
Acute graft versus host disease in liver (Immune system disorders) | 0 | 1
Acute graft versus host disease in skin (Immune system disorders) | 0 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 | 0
Graft versus host disease in liver (Immune system disorders) | 1 | 0
Graft versus host disease in skin (Immune system disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 2 | 0
Heart transplant rejection (Immune system disorders) | 1 | 0
Blastocystis infection (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 3
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Drug level decreased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anosmia (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
Urethral pain (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Blood cholesterol (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT03672292/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT03672292/SAP_001.pdf